CLINICAL TRIAL: NCT06769958
Title: The Effect of Reflexology on Pain, Comfort and Breastfeeding Self-Efficacy in Post-Cesarean Headache Due to Spinal Anesthesia
Brief Title: The Effect of Reflexology on Pain, Comfort and Breastfeeding Self-Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Veysel Can, Asst. Prof., Yuzuncu Yil University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: Reflexology
Record Dates: First submitted 2024-12-31; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Reflexology
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reflexology (Experimental)
  Interventions: Behavioral: Reflexology
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Reflexology — Reflexology application
  Arms: Reflexology

SUMMARY:
This study was conducted to determine the effects of reflexology applied to mothers with headache due to spinal anesthesia after Cesarean delivery on pain, comfort and breastfeeding self-efficacy levels. The study, which was conducted with a single-blind, randomized controlled experimental design, was conducted between April 2024 and August 2024 at the Department of Obstetrics and Pediatrics, SBU Van Training and Research Hospital with mothers who had cesarean delivery under spinal anesthesia and had postpartum headache (Intervention group=30, Control group=30). Foot reflexology was applied to the mothers in the intervention group for a total of 30 minutes, 15 minutes on each foot. The control group was not subjected to any intervention other than routine nursing practices. Personal Information Form, Visual Analog Scale (VAS), Postpartum Comfort Scale (PPSC) and Breastfeeding Self-Efficacy Scale (BSSE) were used as data collection tools.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older,
* performing SD under spinal anesthesia,
* experiencing postpartum headaches,
* Caesarean section performed at 37-42 weeks of gestation,
* giving only one live birth,
* open to written or oral communication,
* at least a primary school graduate,
* no complications during pregnancy,
* mothers who agreed to participate in the study

Exclusion Criteria:

* Performing a cesarean section at periods other than 37-42 weeks of gestation,
* caesarean section under general anesthesia,
* have health problems such as fractures, dislocations, phlebitis, arthritis, burns, wounds, eczema, fungus or inflammation in the foot tissue,
* with disease of the cardiovascular system,
* with chronic diseases such as hypertension or diabetes mellitus,
* Postpartum controlled analgesia administered,
* mothers with psychiatric diagnoses such as anxiety and depression

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | pre-test post-test (approximately eight months), reduce pain
  min-max (0-10), an increased score is a bad result
Postpartum Comfort Scale | pre-test post-test (approximately eight months), Increasing Postpartum Comfort
  min-max (34-170), increased score is a good result
Breastfeeding Self-Efficacy Scale | pre-test post-test (approximately eight months), Increasing breastfeeding self-efficacy
  min-max (14-70), increased score is a good result

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yüzüncü Yıl University, Van, Tuşba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No